CLINICAL TRIAL: NCT03336879
Title: Exploring the Potential of High-frequency Repetitive Transcranial Magnetic Stimulation (rTMS) to Treat Gambling Disorder (GD)
Brief Title: Repetitive Transcranial Magnetic Stimulation in Gambling Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: ITAB - Institute for Advanced Biomedical Technologies (Other)
Responsible Party: Principal Investigator, Giovanni Martinotti, Researcher, ITAB - Institute for Advanced Biomedical Technologies
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: v.2_19/10/2017
Record Dates: First submitted 2017-11-06; First posted 2017-11-08 (Actual); Last update posted 2017-11-08 (Actual); Status verified 2017-11

CONDITIONS: Gambling Disorder
Keywords: Gambling Disorder; Mental Disorder; Behavioral Addiction
MeSH Terms: conditions — Gambling; Mental Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: non-randomized, open label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Active rTMS (15 Hz) (Experimental): The intervention will be Repetitive Transcranial Magnetic Stimulation. Each patient will receive active stimulation targeting the left dorsolateral prefrontal cortex (lDLPFC) with a frequency of 15 Hz and 100% of the individual resting motor threshold, for a total of 40 trains (60 stimuli per train, inter-train interval of 15 second, total duration 13 minutes). Each session will be repeated twice/daily for 10 consecutive days for 2 weeks, during the continued treatment phase. Following this, the participants will receive the maintenance intervention of 2 sessions per week for 3 months (rTMS follow-up), at the same parameters described above. Device: MagPro R30 with the Cool-B80 figure-of-eight coil (MagVenture, Falun, Denmark).
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — Repetitive Transcranial Magnetic Stimulation (rTMS) is a non-invasive brain stimulation technique. The investigators will use a MagPro R30 with the Cool-B80 figure-of-eight coil (MagVenture, Falun, Denmark).
  Other Names: rTMS

SUMMARY:
Background: An imbalance between prefrontal cortex (PFC) and the mesolimbic reward system has been suggested to contribute to GD. GD patients showed increased functional connectivity between regions of the PFC and mesolimbic reward system, as well as reduced connectivity in the area of the PFC. The altered interaction between prefrontal structures and the mesolimbic reward system in GD shares similarity with functional organization reported in Substances Use Disorders (SUDs), suggesting a more general pathophysiology for addictive disorders

Objectives: To test if rTMS can reduce craving and playing in Gambling Disorder, and also affect several mood, behavioral and cognitive alterations associated with prolonged Gambling Disorder.

Eligibility: Healthy, right-handed adults ages 18-65 who do have Gambling Disorder.

Design: This is a non-randomized, open label study. The study includes three phases: 1) a rTMS continued treatment phase; 2) a rTMS follow-up; and 3) a no rTMS follow-up.

Prior to participating, participants will be screened with:

* Questionnaires
* Cognitive tests
* Medical history
* Physical exam

After being enrolled, baseline behavioral and imaging data will be collected. In particular, participants will undergo:

* Questionnaires
* Cognitive tests

During the continued rTMS phase, participants with Gambling Disorder will receive real rTMS. Repetitive TMS will be delivered during 10 outpatient treatment days, over 2 weeks (5 days/week). Following this phase, subjects will have 12 follow-up visits (once/weekly), during which they will receive rTMS, and behavioral assessments will be performed. At the end of the rTMS follow up period, participants will further receive 3 follow up visits (once a month), during which rTMS will not be performed, but behavioral data will be collected.

Treatment includes:

* rTMS: A coil is placed on the head. Brief electrical current passes through the coil. At each visit, participants will receive two rTMS sessions, with a 1hr interval between sessions. At the beginning of each rTMS session, they view gambling-related images for few minutes.
* Repeat of screening tests and questionnaires

DETAILED DESCRIPTION:
Gambling Disorder (GD) is a complex addictive disorder involving fronto-striatal connectivity and prefrontal top-down control modulation of reward-related brain areas. Repetitive transcranial magnetic stimulation (rTMS) seems to reduce cravings and improve cognitive function in substance dependent individuals. Moreover, rTMS has been shown to modulate dopaminergic and glutamatergic transmission, both involved in GD pathophysiology. However, the efficacy of rTMS in treating GD has not been evaluated and also, we lack a full characterization of rTMS effects on other important aspects, including effects on mood, cognition and changes in brain function. The purpose of this study is to investigate the effects of repetitive Transcranial Magnetic Stimulation (rTMS) at 15 Hz frequency on the left dorsolateral prefrontal cortex in patients affected by GD and to examine possible changes in mood, cognition, and brain activity and functional connectivity associated with this intervention. For this purpose, the investigators will recruit GD patients. After screening and informed consent, participants will undergo active rTMS for two consecutive weeks (twice a day) during the continued treatment phase, and a maintenance intervention (twice a week for 3 months), during the rTMS follow-up phase. Following this phase, participants will be followed for further 3 months, during which no rTMS will be delivered but clinical data will be collected.

Procedure: The project consists of: Screening Visit (baseline), Phase 1 (continued treatment phase), Phase 2 (3 months- rTMS follow-up), Phase 3 (3 months follow-up without rTMS). First, there will be a screening visit, where a clinical interview will be conducted and questionnaires and tests will be administered to identify study participants who meet the inclusion and exclusion criteria. Baseline clinical and cognitive data will be acquired. In Phase 1, participants will receive 2 sessions of rTMS (active), twice per day for 10 consecutive days, for a total of 20 rTMS sessions. Following this, the investigators will evaluate the acute effect of treatment on relapse rate, gambling severity and craving, mood and cognition. In Phase 2 of the study, all participants will continue the treatment arm with rTMS (15Hz) for three months. Participants will receive 2 sessions of rTMS (active) once per week; clinical and cognitive data will be acquired once per month. The investigators will evaluate the acute effect of treatment on relapse rate, gambling severity and craving, mood and cognition. In Phase 3 of the study, participants will not receive any rTMS session. Clinical and cognitive data will be acquired once per month for three months. The investigators will evaluate the long-term effect of treatment on relapse rate, gambling severity and craving, mood and cognition.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 65;
* Current diagnosis of Gambling Disorder, based on the Diagnostic and Statistical Manual of Mental Disorder - Fifth Edition (DSM-5);
* Drug-free.

Exclusion Criteria:

* Current DSM-V diagnosis of substance use disorders other than nicotine dependence;
* Current DSM-V diagnosis of schizophrenia, bipolar disorder, or other psychotic disorder;
* Use in the past 4 weeks of any medication with known pro-convulsant action; or current regular use of any psychotropic medications (benzodiazepines, antipsychotic medications, tricyclic antidepressants, anti-epileptics, mood stabilizers);
* Any history of any clinically significant neurological disorder, including organic brain disease, epilepsy, stroke, brain lesions, multiple sclerosis, previous neurosurgery, or personal history of head trauma that resulted in loss of consciousness for > 5 minutes and retrograde amnesia for > 30 minutes;
* Any personal or family history (1st degree relatives) of seizures other than febrile childhood seizures;
* Any psychiatric, medical or social condition whether or not listed above, due to which, in the judgment of the PI and after any consults if indicated, participation in the study is not in the best interest of the patient;
* For female patients: Pregnancy/breastfeeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-12-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Changes in the Visual Analogue Scale for Craving (VAS-craving) | Baseline, after rTMS treatment: 2 weeks, 3 months, 6 months
  A Visual Analogue Scale (VAS) is an instrument to measure a characteristic or attitude that is believed to range across a continuum of values. The VAS is a horizontal line, 100 mm in length, anchored by word descriptors at each end (0 = lower scores; 10 = higher scores). The patient marks on the line the point that they feel represents their perception of their current state. The VAS score is determined by measuring in millimeters from the left-hand end of the line to the point that the patient marks.
Changes in the Pathological Gambling Adaptation of the Yale-Brown Obsessive-Compulsive Scale (PG-YBOCS) | Baseline, after rTMS treatment: 2 weeks, 3 months, 6 months
  The Pathological Gambling Adaptation of the Yale-Brown Obsessive-Compulsive Scale (PG-YBOCS) is a 10-item clinician-administered questionnaire that measures the severity of PG over the past one week. Scores from 0 (min) to 4 (max) are assigned according to the severity. The first set of questions (questions 1-5) assess urges and thoughts associated with pathological gambling, whereas the last five questions assess the behavioral component of the disorder. Both single set scores and total score will be calculated.
Changes in Gambling Disorder Severity as assessed by Timeline Follow Back (TLFB) | Baseline, after rTMS treatment: 2 weeks, 3 months, 6 months, 12 months
  Gambling behavior will be assessed using the TimeLine Follow Back (TLFB). TLFB is an interview-based assessment. Using a calendar, participants are guided through the process of recalling and reporting daily gambling behavior. TLFB provides measures of gambling episodes per week, gambling days per week, heavy gambling days per week.
Changes in Gambling Behavior as assessed by Gambling Symptom Assessment Scale (G-SAS) Total Score | Baseline, after rTMS treatment: 2 weeks, 3 months, 6 months, 12 months
  Gambling Symptom Assessment Scale (G-SAS) is a 12-item self-rated scale designed to assess gambling symptom severity and change during treatment. Each 12-item scale has a score ranging from 0 - 4 (adjective anchors for 0 and 4 vary for each item). All items ask for an average symptom based on the past 7 days. Total score ranges from 0 (min) to 48 (max), higher scores indicate higher severity levels.

SECONDARY OUTCOMES:
Changes in the Iowa Gambling Task (IGT) Performance | Baseline, after rTMS treatment: 2 weeks, 3 months, 6 months
  The Iowa Gambling Task is a computerized card game commonly used to measure risky decision-making tendencies and sensitivity to reward and loss. Performance is calculated on the total net score results from the subtraction of the disadvantageous deck choices from the advantageous deck choices during the entire test ([C'+D']-[A'+B']).
Changes in Snaith Hamilton Pleasure Scale (SHAPS) Total Score | Baseline, after rTMS treatment: 2 weeks, 3 months, 6 months
  The Snaith Hamilton Pleasure Scale (SHAPS) is a 14-item self-report scale designed to measure hedonic-tone/anhedonia. Each item is scored on a 4-point scale, ranging from 0 (not at all) to 3 (extremely). Sum the scores from all 14 parameters gives the SHAPS Total Score which may range from 0 (min) to 42 (max).
Changes in Temporal experience of Pleasure Scale (TEPS) Total | Baseline, after rTMS treatment: 2 weeks, 3 months, 6 months
  The Temporal experience of Pleasure Scale (TEPS) is a 18-item self-report scale designed to evaluate individual trait dispositions in anticipatory and consummatory pleasure experiences. Each item is scored on a 6-point scale, ranging from 1 (extremely false) to 6 (extremely true). Sum the scores from all 20 parameters gives the TEPS Total Score which may range from 20 (min) to 108 (max).
Changes in Montgomery-Asberg Depression Scale (MADRS) Total | Baseline, after rTMS treatment: 2 weeks, 3 months, 6 months]
  The MADRS is a 10-item scale that evaluates the core symptoms and cognitive features of clinical depression. Each MADRS item is rated on a 0 to 6 scale. The MADRS Total score ranges from 0 (min) to 60 (max). Higher MADRS scores indicate higher levels of depressive symptoms.
Changes in Hamilton Rating Scale for Anxiety (HAM-A) Total | Baseline, after rTMS treatment: 2 weeks, 3 months, 6 months
  The HAM-A is a 14-item scale that assesses anxiety symptoms of anxiety such as "anxious mood", "tension" or "fears". Each item is scored on a 5-point scale, ranging from 0 (not present) to 4 (severe). Sum the scores from all 14 parameters gives the HAM-A Total Score which may range from 0 (min) to 56 (max).
Changes in Profile of Mood States (POMS), Total Mood Disturbance Score | Baseline, after rTMS treatment: 2 weeks, 3 months, 6 months
  The profile of mood state (POMS) is a questionnaire designed to measure present mood state by a list of adjectives on a 5-point Likert scale (0 = not at all; 4 = Extremely) and measures six dimensions of affect, including tension-anxiety, depression-dejection, anger-hostility, vigor-activity, fatigue-inertia, and confusion-bewilderment. The measure has been shown to produce reliable and valid profiles of mood state. A Total Mood Disturbance Score may be calculated by adding the scores for Tension, Depression, Anger, Fatigue and Confusion and then subtracting the score for Vigor.

CONTACTS AND LOCATIONS:
Overall Officials: Massimo di Giannantonio, MD, Principal Investigator — Department of Neuroscience, Imaging and Clinical Sciences (ITAB) - University G. d'Annunzio - Chieti (Italy)
Locations (2):
- Italy (2):
  - Department of Neuroscience, Imaging and Clinical Sciences, Chieti
  - La Promessa ONLUS, Roma

REFERENCES:
- [Derived] Pettorruso M, Martinotti G, Montemitro C, De Risio L, Spagnolo PA, Gallimberti L, Fanella F, Bonci A, Di Giannantonio M; Brainswitch Study Group. Multiple Sessions of High-Frequency Repetitive Transcranial Magnetic Stimulation as a Potential Treatment for Gambling Addiction: A 3-Month, Feasibility Study. Eur Addict Res. 2020;26(1):52-56. doi: 10.1159/000504169. Epub 2019 Oct 30. PMID 31665732

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-19): https://cdn.clinicaltrials.gov/large-docs/79/NCT03336879/Prot_SAP_000.pdf